CLINICAL TRIAL: NCT00619879
Title: Myeloablative Hematopoietic Progenitor Cell Transplantation (HPCT) for Pediatric Malignancies
Status: Completed | Type: Observational
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Sonali Chaudhury, MD, Principal Investigator, Ann & Robert H Lurie Children's Hospital of Chicago
Other Study IDs: SCT 0307
Record Dates: First submitted 2008-01-08; First posted 2008-02-21 (Estimated); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Leukemia, Myelogenous, Chronic; Leukemia, Lymphoblastic, Acute; Leukemia, Myelogenous, Acute; Myeloproliferative-Myelodysplastic Diseases; Lymphoma, Malignant
Keywords: Leukemia, Myelogenous, Chronic; Leukemia, Lymphoblastic, Acute; Leukemia, Myelogenous, Acute; Myeloproliferative-Myelodysplastic Diseases; Juvenile Myelomonocytic Leukemia; Dysmyelopoietic Syndromes; Lymphoma, Malignant; Stem Cell Transplantation, Hematopoietic; Allogeneic Transplantation; Human Leukocyte Antigens; Busulfan; Total Body Irradiation; VP-16; Etoposide; Cyclophosphamide; Graft-Versus-Host Disease
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Myelodysplastic-Myeloproliferative Diseases; Lymphoma; Leukemia, Myelomonocytic, Juvenile; Myelodysplastic Syndromes; Graft vs Host Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Myeloablative Chemotherapy Regimen for Lymphoid Malignancies or Cord Blood Unit Recipients — Total Body Irradiation (TBI) 1200 cGy will be given on days -8,-7,-6 and -5 in eight sessions, delivering 150cGy in each session.
  Etoposide 1000 mg/m2 as a 24 hour continuous infusion started on day -4.
  Cyclophosphamide 60 mg/kg/day IV given over 1 hour daily on days -3, -2.
Drug: Myeloablative Chemotherapy Regimen for Non-Cord Blood Unit Recipients with Myeloid Malignancies — Busulfan administration:
  * For children >/= 4 years of age, Busulfan 0.8 mg/kg/dose will be given every 6 hours over days -8,-7, -6, and -5 for a total of 16 doses.
  * For children < 4 years of age, Busulfan 1 mg/kg/dose will be given every 6 hours over days -8, -7, -6, -5 for a total of 16 doses.
  * Pharmacokinetic analysis will guide dose modifications targeted to receive an average AUC of 800-1200 microMols*min for the 16 doses.
  Lorazepam (0.05 mg/kg) IV will be administered one half hour before the initial dose of Busulfan is given and every 6 hours through day -4.
  Etoposide 1000 mg/m2 as a 24 hour continuous infusion started on day -4.
  Cyclophosphamide 60 mg/kg/day IV given over 1 hour daily on days -3 and -2.
Other: Hematopoietic Progenitor Cell Transplantation (HPCT) — Hematopoietic progenitor cells (HPCs) will be infused on day 0. Source of cells may be bone marrow, peripheral blood cells, or cord blood units, from matched related or unrelated donors.
Radiation: CNS radiation treatment for ALL with prior CNS disease patients — Patients with prior CNS disease over the age of 1 year will be treated with 600 cGy of cranial irradiation in addition to 1200 cGy of TBI.
  Patients diagnosed with ALL with CNS disease (at the time of diagnosis or relapse) < 1 year of age will receive CNS treatment as Intrathecal Methotrexate as follows:
  * Infants ≤ 1 year of age at the time of Intrathecal Therapy will receive a dosing of 7.5 mg once a month for 6 months after transplant beginning at day +30 with an adequate white count
  * Children 1-2 years of age at the time of Intrathecal Therapy will receive 8 mg once a month for 6 months after transplant beginning at day +30 with an adequate white count

SUMMARY:
The purpose of this study is to show that myeloablative hematopoietic progenitor cell transplantation (HPCT) continues to offer acceptable disease-free survival for select patients requiring HPCT.

DETAILED DESCRIPTION:
Myeloablative hematopoietic progenitor cell transplantation (HPCT) remains the standard of care for patients requiring HPCT. The purpose of this study is to evaluate the morbidity and mortality of myeloablative HPCT at Children's Memorial Hospital. It will also look to determine the toxicity of a single conditioning regimen consisting of total body irradiation (TBI), etoposide (VP-16), and Cyclophosphamide for patients with transplant eligible lymphoid malignant conditions or with transplant eligible myeloid malignant conditions who are receiving cord blood units, or to determine the toxicity of a single conditioning regimen consisting of Busulfan and Cyclophosphamide for patients with transplant eligible myeloid malignant conditions who are not receiving cord blood units.

ELIGIBILITY:
Inclusion Criteria:

* Malignant Disease

  * Chronic myleogenous leukemia in chronic or accelerated phase
  * Acute lymphoblastic leukemia (ALL)

    * First remission high-risk ALL (Ph+, t( 4-11) infants).
    * Second remission ALL, after a short first remission (<36 mos from Dx).
    * 3rd or greater remission ALL.
  * Acute myelogenous leukemia (AML)

    * First remission high risk acute nonlymphoblastic (ANLL) (as defined by cytogenetics), if a matched sibling donor is available.
    * Initial partial remission AML (<20% blasts in the bone marrow).
    * AML that is refractory to two cycles of induction therapy.
    * Second or greater remission AML
  * Myelodysplastic/Myeloproliferative Disease

    * Juvenile Myelomonocytic Leukemia (JMML)
    * Myelosplastic syndrome and/or pre-leukemia at any stage
  * Lymphoma

    * Relapsed lymphoma with residual disease that appears to be chemo-sensitive and non-bulky (<5 cm at largest diameter)
* Venous Access: Three lumens of central vascular access will be required for all patients entered on protocol due to the need for a dedicated line for continuous infusion cyclosporine.
* Informed Consent: The patient and/or the patient's legally authorized guardian must acknowledge in writing that consent to become a study subject has been obtained in accordance with the institutional policies approved by the U.S. Department of Health and Human Services.
* Patient organ function requirements:

  * Adequate renal function: Serum Creatinine <~1.5 x normal, or Creatinine clearance of 70 mL/min/1.73 mE2 or an equivalent GFR as determined by the institutional normal range
  * Adequate liver function: Total bilirubin <1.5 x normal; and SGOT (AST) or SGPT (ALT) <~2.5 x normal
  * Adequate cardiac function: Shortening fraction of >/=27% by echocardiogram
  * Adequate pulmonary function: FEV1/FVC >/=60% by pulmonary function test; for children who are uncooperative, no evidence of dysnpea at rest, or exercise intolerance, and must have a pulse oximetry >94% in room air
* Performance status: Lansky for children </= 16 years >/= 60; Karnofsky status for those > 16 years of age >/= 70
* Effective Contraceptive Use: Women of childbearing potential and sexually active males should use effective contraception while on study.

Exclusion Criteria:

* Patients who are pregnant or lactating
* Inability to find a suitable donor for the patient
* Patient is HIV-positive
* Patient has active Hepatitis B
* Disease progression or relapse prior to HPC infusion

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients that meet the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2007-03-26 (Actual); Primary Completion 2019-02-07 (Actual); Study Completion 2019-02-07 (Actual)

PRIMARY OUTCOMES:
Evaluate the morbidity and mortality of hematopoietic progenitor cell transplantation (HPCT) at Children's Memorial Hospital. | To study end

SECONDARY OUTCOMES:
Evaluate the effectiveness of graft versus host disease prevention with a combination of anti-thymocyte globulin, continuous infusion cyclosporine, and short course methotrexate for transplants. | To study end
Determine the toxicity of a single conditioning regimen consisting of total body irradiation, etoposide, and Cyclophosphamide for patients with transplant eligible lymphoid malignant conditions or myeloid malignant conditions receiving cord blood units. | To study end
Determine the toxicity of a single conditioning regimen consisting of Busulfan and Cyclophosphamide for patients with transplant eligible myeloid malignant conditions who are not receiving cord blood units. | To study end

CONTACTS AND LOCATIONS:
Overall Officials: Sonali Chaudhury, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States